CLINICAL TRIAL: NCT02251925
Title: Comparison of Pregnancy Outcomes in Frozen Embryo Transfer in Natural and Hormonal Replacement Cycles: a Randomized Controlled Trial
Brief Title: Frozen Embryo Transfer in Natural and Hormonal Replacement Cycles
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-019
Record Dates: First submitted 2014-09-23; First posted 2014-09-29 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2012-04

CONDITIONS: Infertility
Keywords: infertility froze emberyo transfer hormone replacement
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Natural cycle (Experimental): In natural cycle without hCG, daily monitoring of urinary LH is started from day eight of the cycle and frozen-thawed embryo transfer is planned 3-5 days after detection of LH surge, observing mature follicles in ultrasound and endometrial thickness over 7mm for cleavage embryos.
  Interventions: Biological: frozen Embryo transfer
- Natural cycle + hCG for ovulation induction (Experimental): In natural cycle with hCG, after detection of mature follicles in ultrasound and endometrial thickness over 7mm, 10,000IU hCG is injected for ovulation and embryo transfer is performed 3-5 days later in cleavage stage.
  Interventions: Biological: frozen Embryo transfer; Drug: 10,000U hCG injection
- Hormonally controlled cycle with GnRH-a (Experimental): In this group , injection of GnRH agonist (Superfact) at a subcutaneous daily dose of 0.5 mg is started on the day 17-19 of the natural menstrual cycle. Once pituitary desensitization is confirmed, hormonal treatment is commenced with 4mg/day oral Estradiol valerate and after 7 days if endometrial thickness is adequate, Estradiol administration will be continued with the same dose and 100mg Progesterone is administered before embryo transfer, otherwise patients are candidates for higher dosage of Estradiol till favourable endometrial thickness is achieved.
  Interventions: Biological: frozen Embryo transfer; Drug: GnRH agonist (Superfact)
- Hormonally controlled cycle without GnRH-a (Experimental): In the hormonal group without GnRH-a, endometrial preparation will be started with daily administration of 6 mg Estradiol valerate from the 2nd day of the natural menstrual cycle for 6 days. Then treatment will be continued similar to the 3rd group.
  Interventions: Biological: frozen Embryo transfer; Drug: administration of 6 mg Estradiol valerate

INTERVENTIONS:
Biological: frozen Embryo transfer — In this study all patients who will undergo frozen embryo transfer are randomly allocated to be prepared for transfer by using either natural cycle (with or without hCG for ovulation induction) or Hormonal cycle (with or without administration of GnRH-a).
Drug: 10,000U hCG injection — In natural cycle with hCG, after detection of mature follicles in ultrasound and endometrial thickness over 7mm, 10,000IU hCG is injected for ovulation and embryo transfer is performed 3-5 days later in cleavage stage.
  Arms: Natural cycle + hCG for ovulation induction
Drug: GnRH agonist (Superfact) — In group 3, injection of GnRH agonist (Superfact) at a subcutaneous daily dose of 0.5 mg is started on the day 17-19 of the natural menstrual cycle. Once pituitary desensitization is confirmed, hormonal treatment is commenced with 4mg/day oral Estradiol valerate and after 7 days if endometrial thickness is adequate, Estradiol administration will be continued with the same dose and 100mg Progesterone is administered before embryo transfer, otherwise patients are candidates for higher dosage of Estradiol till favourable endometrial thickness is achieved.
  Arms: Hormonally controlled cycle with GnRH-a
Drug: administration of 6 mg Estradiol valerate — In the hormonal group without GnRH-a, endometrial preparation will be started with daily administration of 6 mg Estradiol valerate from the 2nd day of the natural menstrual cycle for 6 days. Then treatment will be continued similar to the 3rd group.
  Arms: Hormonally controlled cycle without GnRH-a

SUMMARY:
This study is a prospective randomized controlled trial to compare the pregnancy outcomes of frozen embryo transfer in natural and hormonal replacement cycles. The study population consisted of all infertile women with regular menstrual cycles who will undergo IVF/ICSI and frozen embryo transfer in Reproductive Biomedicine Research Center, Royan institute, Tehran Iran.

DETAILED DESCRIPTION:
In this study all patients who will undergo frozen embryo transfer are randomly allocated to be prepared for transfer by using either natural cycle (with or without hCG for ovulation induction) or Hormonal cycle (with or without administration of GnRH-a) In natural cycle without hCG, daily monitoring of urinary LH is started from day eight of the cycle and frozen-thawed embryo transfer is planned 3-5 days after detection of LH surge, observing mature follicles in ultrasound and endometrial thickness over 7mm for cleavage embryos.

In natural cycle with hCG, after detection of mature follicles in ultrasound and endometrial thickness over 7mm, 10,000IU hCG is injected for ovulation and embryo transfer is performed 3-5 days later in cleavage stage.

In group 3, injection of GnRH agonist (Superfact) at a subcutaneous daily dose of 0.5 mg is started on the day 17-19 of the natural menstrual cycle. Once pituitary desensitization is confirmed, hormonal treatment is commenced with 4mg/day oral Estradiol valerate and after 7 days if endometrial thickness is adequate, Estradiol administration will be continued with the same dose and 100mg Progesterone is administered before embryo transfer, otherwise patients are candidates for higher dosage of Estradiol till favourable endometrial thickness is achieved.

In the hormonal group without GnRH-a, endometrial preparation will be started with daily administration of 6 mg Estradiol valerate from the 2nd day of the natural menstrual cycle for 6 days. Then treatment will be continued similar to the 3rd group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with regular mensturation cycles
2. Age 20-37 years
3. Patients who underwent long protocol
4. Body mass index (BMI) ≤ 30 kg/m2
5. Patients who will undergo frozen embryo transfer for the first time

Exclusion Criteria:

1. Oocyte or embryo donation cycles
2. Uterine diseases or malformations
3. Hyper prolactinemia
4. Thyroid disorders
5. Tuberculosis
6. Recurrent abortion history
7. Severe endometriosis
8. Ovulation disorders

Ages: 20 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 460 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks
  The pregnancy rate will be evaluated in patients of each groups 4-6 weeks after embryo transfer.

SECONDARY OUTCOMES:
Implantation rate | 4 weeks
  Evaluation the implantation rate in patients of each groups 4-6 weeks after frozen embryo transfer
chemical pregnancy rates | 2 weeks
  Evaluation the chemical pregnancy rates in patients of each group 2 weeks after embryo transfer.
Ongoing pregnancy | 12 weeks
  Evaluation the ongoing pregnancy in patients of each group 12 weeks after embryo transfer.
miscarriage rate | 12 weeks
  Evaluation the miscarriage rate in patients of each group 12 weeks after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Tahereh Madani, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran; Ladan Mohammadi Yeganeh, MSC, Principal Investigator — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Madani T, Ramezanali F, Yahyaei A, Hasani F, Bagheri Lankarani N, Mohammadi Yeganeh L. Live birth rates after different endometrial preparation methods in frozen cleavage-stage embryo transfer cycles: a randomized controlled trial. Arch Gynecol Obstet. 2019 Apr;299(4):1185-1191. doi: 10.1007/s00404-019-05062-7. Epub 2019 Feb 1. PMID 30707360
- See also: Related Info — http://Royaninstitute.org